CLINICAL TRIAL: NCT04331171
Title: Epidemiological Observation From a Smartphone Self-monitoring Application for Suspected COVID-19 Patients' Triage
Acronym: COVID CALL 15
Status: Completed | Type: Observational
Sponsor: Weprom (Other)
Collaborators: Institut Pasteur (Industry); Assistance Publique - Hôpitaux de Paris (Other); DOCAPOST (Unknown); Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Other Study IDs: WP-2020-02
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: COVID-19
Keywords: M-health; COVID-19; Self-assessment application; epidemiology; symptoms
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Web-application users: questionnaire of comorbidity and symptomes completed by the user on his smartphone
  Interventions: Device: Web application users

INTERVENTIONS:
Device: Web application users — questionnaire of comorbidity and symptoms completed by the patient on his smartphone

SUMMARY:
A coronavirus pandemic began on 12/31/2020 with the first Chinese patient. As of 3/16/2020, the epidemic affects more than 100 countries with 169,000 official infections and 6,500 deaths. This virus causes a pathology ranging from simple flu symptoms in 80% of cases to acute respiratory distress syndromes requiring resuscitation in 5% of cases and a death rate of 1.4 to 4% of cases.

The arrival in France on 02/25/2020 with an exponential development of the infection (more than 5,000 cases on 03/15/2020) was accompanied by an unprecedented number of calls to the French emergency service call number (15) of worried patients with overload and sometimes saturation of the service that can impact calls and the care of patients really recovering from an emergency.

We previously developed a Moovcare® web application which showed a 7 months survival benefit by early detection of relapsed lung cancer based on the reporting of patient symptoms analyzed by a validated algorithm in 300 patients and 1 trial randomized. Another application for detecting and monitoring chemo-induced febrile aplasia appears to show a reduction in the number of hospitalizations for sepsis. Finally, Smokecheck, a self-assessment application for symptoms by smokers, has shown that it improves the detection of symptomatic operable bronchial cancers (9 to 24%, p = 0.04).

The web application https://www.maladiecoronavirus.fr/ was developed with a group of physicians from the Institut Pasteur, Hospitals group of Paris, Hospitals of Lille and Rennes and the ILC Jean Bernard in Le Mans. It makes it possible to guide symptomatic patients and patients who wishing to know what to do (call their general practitioner, teleconsultation, or call emergency service) based on symptoms and predictive factors of severity.

Following the availability of this new tool, we want to assess the impact of the application on the number and relevance of calls to emergency service.

ELIGIBILITY:
Inclusion Criteria:

* All users of the https://www.maladiecoronavirus.fr/ application over the age of 18

Exclusion Criteria:

* not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All users of the https://www.maladiecoronavirus.fr/ application over the age of 18
Sampling Method: Probability Sample
Enrollment: 12000000 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
To assess of the evolution of the number of calls to Emergency service within 12 days after the launch of the application https://www.maladiecoronavirus.fr/ | 12 days
  Number of calls to Emergency service after the launch of web application comparded to the days before
To assess of the evolution of the proportion of relevant calls to Emergency service within 12 days after the launch of the application https://www.maladiecoronavirus.fr/ | 12 days
  Number of relevants calls to Emergency service after the launch of web application comparded to the days before

SECONDARY OUTCOMES:
To assess the evolution over time of the COVID 19 epidemic | 3 months
  the symptoms collected by the application
To assess the evolution over space of the COVID 19 epidemic | 3 months
  the symptoms collected by the application according to ZIP code
To assess symptoms | 3 months
  Descriptive analysis of symptoms collected by web-application
To assess the users population | 3 months
  Descriptive analysis of data collected by web-application

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice DENIS, MD, Study Director — Jean Bernard Center - LE MANS
Locations (1):
- All French Emergency services, Le Mans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Denis F, Fontanet A, Le Douarin YM, Le Goff F, Jeanneau S, Lescure FX. A Self-Assessment Web-Based App to Assess Trends of the COVID-19 Pandemic in France: Observational Study. J Med Internet Res. 2021 Mar 12;23(3):e26182. doi: 10.2196/26182. PMID 33709945
- [Derived] Galmiche S, Rahbe E, Fontanet A, Dinh A, Benezit F, Lescure FX, Denis F. Implementation of a Self-Triage Web Application for Suspected COVID-19 and Its Impact on Emergency Call Centers: Observational Study. J Med Internet Res. 2020 Nov 23;22(11):e22924. doi: 10.2196/22924. PMID 33147165
- [Derived] Denis F, Galmiche S, Dinh A, Fontanet A, Scherpereel A, Benezit F, Lescure FX. Epidemiological Observations on the Association Between Anosmia and COVID-19 Infection: Analysis of Data From a Self-Assessment Web Application. J Med Internet Res. 2020 Jun 11;22(6):e19855. doi: 10.2196/19855. PMID 32496206